CLINICAL TRIAL: NCT02215343
Title: Effect of Prebiotic Fibre and Polyunsaturated Fatty Acid (PUFA) on the Gut Microbiota and Metabolic Risk Markers in a Metabolically Challenged Population
Brief Title: Effect of Prebiotic and PUFA on the Gut Microbiota and Metabolic Risk Markers
Acronym: MyNewGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: http://mynewgut.eu/partners (Unknown)
Responsible Party: Principal Investigator, Arne Astrup, Professor, Dr.Med., University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MyNewGut, Task 3.3; Grant Agreement no: 613979 (Other Grant/Funding Number: EU 7th Framework Programme)
Record Dates: First submitted 2014-07-15; First posted 2014-08-13 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Dietary Fiber; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High fibre diet (wheat bran extract) (Experimental)
  Interventions: Dietary Supplement: Wheat bran extract
- High PUFA diet (fish oil supplement) (Experimental)
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Wheat bran extract — Patients will be provided with 15g of wheat bran extract (WBE) (Cargill R&D Centre Europe).
  Arms: High fibre diet (wheat bran extract)
Dietary Supplement: Fish oil — Patients will be provided with a fish oil supplement (capsules), containing 3-4g of N-3 fatty acids (Axellus A/S, Ishøj, Denmark).
  Arms: High PUFA diet (fish oil supplement)

SUMMARY:
The main objective of this study is to investigate in detail how a high-(prebiotic)fibre diet and a high-PUFA diet affect the gut microbiota composition in a metabolic challenged population, and if the diet-induced modulation of the gut microbiota mediates changes in metabolic risk markers.

Intake of both experimental diets over 4 weeks are expected to induce beneficial changes in the gut microbiota composition and to affect markers for insulin sensitivity, lipid metabolism and inflammation. The investigators hypothesize that the effect of both interventions on the metabolic risk markers will be partly mediated by the diet-induced changes in the gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-40 kg/m2
* Non-smoking
* Indices of the Metabolic Syndrome defined by the International Diabetes Federation (IDF 2006):

Central obesity (waist circumference; men: ≥94 cm and women: ≥80 cm) + any one of the following; raised triglyceride level (≥1.7 mmol/L), reduced HDL cholesterol (men: <1.03 mmol/L, women: <1.29 mmol/L), raised BP (systolic ≥130 mm Hg or diastolic ≥85 mm Hg) or raised fasting plasma glucose (≥5.6 mmol/L).

Exclusion Criteria:

* Use of antibiotics
* Weight change >3 kg 2 months prior to study start
* Intensive physical training/ elite athlete
* Medication for dyslipidemia, type 2 diabetes or elevated blood pressure
* Dietary supplements with pro/prebiotics, dietary fibre or fish oil supplement
* Lactation, pregnancy or planning of pregnancy during the study
* Gastro intestinal and liver disorders
* Chronic inflammatory disorders
* Diagnosed psychiatric disorder including treatment required depression
* Surgical treatment of obesity and abdominal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota composition | Week 0, 4, 8, 12
  Gut microbiota composition will be analyzed by use of fecal samples.

SECONDARY OUTCOMES:
Change in markers for insulin sensitivity | Week 0, 4, 8, 12
  Will be measured by use of fasting blood samples
Change in markers for lipid metabolism | Week 0, 4, 8, 12
  Will be measured by use of fasting blood samples
Change in markers for inflammation | Week 0, 4, 8, 12
  Will be measured by use of fasting blood samples
Faecal SCFA and bile acid composition | Week 0, 4, 8, 12
  Will be analyzed by use of fecal samples.
Lipidomics | Week 0, 4, 8, 12
  Will be analyzed by use of fasting blood samples and fecal samples.
Metabolomics | Week 0, 4, 8, 12
  Will be analyzed by use of fasting blood samples, urine and fecal samples.

OTHER OUTCOMES:
Change in energy expenditure | Week 0, 4, 8, 12
  Resting energy expenditure will be measured by indirect calorimetry in a ventilated hood system
Gene expression | Week 0, 4, 8, 12
  Adipose tissue biopsies will be used for epigenetic analyses, gene and protein expression (no whole genome or exome sequencing).
Compliances markers | Week 0, 4, 8, 12
  Compliance will be evaluated from 3-days diet registration and self-reported intake of dietary supplements, PUFA complance markes (fatty acid composition) and body composition

CONTACTS AND LOCATIONS:
Overall Officials: Lesli H Larsen, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Benitez-Paez A, Kjolbaek L, Gomez Del Pulgar EM, Brahe LK, Astrup A, Matysik S, Schott HF, Krautbauer S, Liebisch G, Boberska J, Claus S, Rampelli S, Brigidi P, Larsen LH, Sanz Y. A Multi-omics Approach to Unraveling the Microbiome-Mediated Effects of Arabinoxylan Oligosaccharides in Overweight Humans. mSystems. 2019 May 28;4(4):e00209-19. doi: 10.1128/mSystems.00209-19. PMID 31138673
- [Derived] Kjolbaek L, Benitez-Paez A, Gomez Del Pulgar EM, Brahe LK, Liebisch G, Matysik S, Rampelli S, Vermeiren J, Brigidi P, Larsen LH, Astrup A, Sanz Y. Arabinoxylan oligosaccharides and polyunsaturated fatty acid effects on gut microbiota and metabolic markers in overweight individuals with signs of metabolic syndrome: A randomized cross-over trial. Clin Nutr. 2020 Jan;39(1):67-79. doi: 10.1016/j.clnu.2019.01.012. Epub 2019 Feb 19. PMID 30827722